CLINICAL TRIAL: NCT04656639
Title: Diffusion-Weighted MRI for Diagnosis of Multifocal, Multicentric Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Kyung Moon, Professor, Seoul National University Hospital
Other Study IDs: 2007-206-1145
Record Dates: First submitted 2020-10-11; First posted 2020-12-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Detection of multifocal, multicentric breast cancer in patients with breast cancer affects surgical decision. Histology-proven additional cancer foci have been reported to be detected in 21.0% to 63.0% of affected breasts in women thought to have localized cancer based on clinical assessment and mammography. Dynamic contrast-enhanced (DCE) MRI is often applied in the preoperative local staging of breast cancer due to its high sensitivity and identifies additional foci that would have otherwise remained undetected on clinical assessment and conventional imaging (mammography and ultrasonography). However, DCE MRI is limited in use due to its low specificity with high false positive rate, causing unnecessary and incorrect conversion to more extensive surgery. Diffusion-weighted MRI (DWI) is a fast, functional MRI technique that measures the movement of water molecules to create tissue contrast without the need for contrast injection. Breast malignancies exhibit hindered diffusion and appear hyperintense on DWI with low apparent diffusion coefficient (ADC) values compared to normal surrounding tissue or benign tumors. Multiple studies including one prospective multi-center trial showed that DWI can reduce unnecessary benign biopsies of suspicious mammographic or DCE MRI-detected lesions and DWI is now considered as an important part of multi-parametric breast MRI protocols. However, little is known about the role of DWI as an adjunct to DCE MRI in the local staging of women with breast cancer. The purpose of our study is to determine whether DWI improves the performance of preoperative DCE MRI in the evaluation of additional lesions in breast cancer patients.

DETAILED DESCRIPTION:
Primary objective: to compare the diagnostic performance of DCE MRI vs combination of DWI and DCE MRI for detection of multifocal, multicentric breast cancer in patients planning for breast conservation surgery

Detailed Description

* This is a multicenter, intraindividual comparative cohort study.
* A total of 580 women with newly diagnosed breast cancer will be enrolled in this study.
* Each eligible woman with newly diagnosed invasive breast cancer will undergo DCE MRI and DWI at a 3T MR scanner.
* Contrast-enhanced MRI and DWI will be interpreted independently according to the Breast Imaging Reporting and Data System (BI-RADS) and likelihood of malignancy (Score range, 0%-100%) by trained radiologists.
* Multifocal breast cancer is defined as presence of more than 2 separate (≥1.0cm) foci of breast cancer in the same quadrant or within 5 cm of the primary lesion.
* Multicentric cancer is defined as two or more synchronous ipsilateral neoplasm located in different quadrant or beyond 5 cm from the primary lesion.
* BI-RADS final assessment score of 4 or 5 are considered to be positive.
* Pathology of core or surgical biopsy and 2 year follow up is the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Women aged more than 25 years at the time of enrollment
* Women underwent digital mammography and whole-breast US before MRI
* Women with image-guided biopsy result of invasive breast cancer
* Women who are planning for breast conservation surgery
* Women who will undergo preoperative breast MRI

Exclusion Criteria:

1. Women aged less than 25 years at the time of enrollment
2. Women with image-guided biopsy result of ductal carcinoma in situ or recurrent breast cancer
3. Women who underwent lumpectomy before MRI
4. Women receiving neoadjuvant chemotherapy or undergoing chemotherapy due to other malignancy
5. Pregnant or lactating women
6. Women with contraindication to breast MRI (claustrophobia, renal insufficiency GFR <60mL/min/1.73m2, metallic foreign body, history of severe side effects due to MR contrast agent, who cannot tolerate 40 minute scanning time etc).

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients planning for breast conservation surgery
Sampling Method: Non-Probability Sample
Enrollment: 580 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Receiver operating characteristic per lesion and breast level | 2 year after enrollment
  Area under the curve (AUC)

SECONDARY OUTCOMES:
Sensitivity per lesion and breast level | 2 year after enrollment
  Number of positive examinations with a tissue diagnosis of cancer within 2 year/All examinations with tissue diagnosis of cancer within the same period
Specificity per lesion and breast level | 2 year after enrollment
  Number of negative examinations without tissue diagnosis of cancer within 2 year/All examinations without tissue diagnosis of cancer within the same period
Positive Predictive value per lesion and breast level | 2 year after enrollment
  True positive/True positive + False positive
Characteristics of detected cancers | 2 year after enrollment
  Tumor size, type, grade, molecular subtype, and lymph node metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Woo Kyung Moon, Study Chair — Seoul National University Hosptial
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park VY, Shin HJ, Kang BJ, Kim MJ, Moon WK, Song SE, Ha SM. Diffusion-Weighted Magnetic Resonance Imaging for Preoperative Evaluation of Patients With Breast Cancer: Protocol of a Prospective, Multicenter, Observational Cohort Study. J Breast Cancer. 2023 Jun;26(3):292-301. doi: 10.4048/jbc.2023.26.e18. Epub 2023 Apr 6. PMID 37272245